CLINICAL TRIAL: NCT02045134
Title: Supplementation With Polyphenol-Rich Foods and Atrial Fibrillation After a Cardiac Surgery
Acronym: Polyphemus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low participation rate
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Licia Iacoviello, Laboratory Head, Neuromed IRCCS
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Neuromed-GR-2008-1146478
Record Dates: First submitted 2014-01-20; First posted 2014-01-24 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2016-07

CONDITIONS: Coronary Heart Disease
Keywords: Post Operative Atrial Fibrillation after a cardiac surgery
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Soluble corn flour not rich in anthocyanins
  Interventions: Dietary Supplement: Placebo
- High-anthocyanin rich corn flour (Active Comparator): Soluble corn flour at high content in anthocyanins
  Interventions: Dietary Supplement: High-anthocyanin rich corn flour

INTERVENTIONS:
Dietary Supplement: Placebo — Soluble corn flour not rich in anthocyanins
  Arms: Placebo
Dietary Supplement: High-anthocyanin rich corn flour — Soluble corn flour at high content in anthocyanins
  Arms: High-anthocyanin rich corn flour

SUMMARY:
Post-operative atrial fibrillation (POAF) is a major cause of morbidity and mortality after a cardiac surgery. Both systemic inflammation and oxidative stress play a role in the initiation of POAF after a cardiac surgery. Epidemiological studies show a significant inverse correlation between cardiovascular risk and consumption of polyphenol-rich foods (PRFs), due to antioxidant, vasorelaxant and antithrombotic properties of their polyphenolic components. The main objective of this study is to evaluate the effect of polyphenol-rich food supplementation on post-operative atrial fibrillation (POAF) in patients undergoing an open heart surgery (mainly coronary artery bypass grafts (CABG) and valve replacement or repaired (VR))

DETAILED DESCRIPTION:
1. Study Rationale: An open heart surgery (OHS) induces injury of the vessel wall and is characterized by post-operative complications. Post-operative atrial fibrillation (POAF) is a major cause of morbidity and mortality after cardiac surgery. Both systemic inflammation and oxidative stress play a role in the initiation of POAF after a cardiac surgery. Consumption of polyphenol-rich foods (PRFs), such as fruits and vegetables, and beverages derived from plants, such as cocoa, red wine and tea, may represent a beneficial diet in terms of cardiovascular protection. Indeed, epidemiological studies demonstrate a significant inverse correlation between PRFs consumption and cardiovascular risk, due to antioxidant, vasorelaxant and antithrombotic properties of their polyphenolic components. In particular, procyanidins from grape seeds are the principal vasoactive polyphenols in red wine and protect endothelial cells from oxidative damage. However, there are no studies that have addressed the relationship of PRFs consumption with prognosis in patients undergoing an OHS.
2. Aim of the study. The main objectives of this project are to evaluate the association between the effect of polyphenol-rich food supplementation and post-operative atrial fibrillation (POAF) in patients undergoing an OHS.
3. Study design: Multicentre, randomized, placebo-controlled double-blind trial with 2 parallel arms: soluble corn flour at high content in anthocyanins and placebo. Placebo consists of soluble corn flour not rich in anthocyanins. The treatment will start at hospital admission until one day before cardiac surgery, and continue (4 days) after extubation and when the patients are reallocated to eat.
4. Study Population and recruitment: A total of 350 consecutive CAD patients undergoing to CABG or VR will be recruited. Participants will be identified at the Department of Cardiovascular disease of the clinical centers.

   Eligible subjects will be recruited at their first surgical consultation and subsequently referred to the research investigators. The research staff in charge of the recruitment will pre-screen participants on the basis of inclusion/exclusion criteria and will explain the study at this time.

   The main inclusion criteria are :age 18 years or older, presence of sinus rhythm on the screening electrocardiogram, first-time elective open heart surgery. Exclusion criteria are: absence of sinus rhythm at screening, known allergy or intolerance to gluten or anthocyanin compound, regularly consuming of anthocyanin or antioxidant supplements, being currently pregnant, existing or planned cardiac transplant or use of ventricular assist device, or being unable or unwilling to provide informed consent, known history of hepatic or renal disease, cancer and subjects with a history of substance abuse.

   Once signed the informed consent, if the subject is eligible for the study according to the inclusion/exclusion criteria, he/she will be included into the trial and randomised, using prepared envelopes blinded to the study investigators, to receive daily high-anthocyanin supplement or placebo.

   Subjects will start the dietary intervention at hospital admission until one day before cardiac surgery. Then they will continue the supplementation as soon they are reallocated to eat for the next 4 days after the surgery.

   Each patient will be asked to answer electronic questionnaires to collect personal information and medical history (social status, previous disease or surgical interventions, risk factors and family history for cardiovascular disease, drug use). Other relevant clinical data as well as measures of clinical outcomes will be collected by medical records. A 1-year food frequency questionnaire will be used to investigate dietary habits. Electrocardiographic, blood pressure, anthropometric measurements will be collected using standardized methods. During the hospitalization, time in intensive therapy, post-surgical course, specific drug therapy, post-surgical complications, fatal and non-fatal cardiovascular events, re-intervention of revascularization and bypass occlusion will be recorded.

   Venous blood (max 30 mL) will be collected before PRFs/placebo supplementation and 24 h and 72 h after the cardiac surgery.

   The patients will undergo OHS according to the indication and good practice procedures normally applied in the Department of Cardio-surgery of participant clinical centers.

   All patients will receive the pharmacological therapy and the lifestyle change advice according to the best clinical practice for the specific disease and surgical intervention.
5. Evaluation criteria: The primary end point will be the occurrence of postoperative AF of at least 30 seconds' duration and documented by rhythm strip or 12-lead ECG or treated with pharmacological or electrical cardioversion.
6. Power calculation: Fixing alpha=0.05, beta=0.2, the incidence of POAF =38% with a sample size of N=350 CABG patients (half of them will be randomize to PRFs supplementation) and a 22% of drop-out, we can observe a relative risk <0.64 in reduction of POAF in the intervention group.
7. Statistical analysis. All analyses will be performed using statistical analysis software SAS (SAS, 9.1.3 for Windows, Cary, NC: SAS Institute Inc.1989). All individuals enrolled will be included in the analysis. Descriptive summaries will be presented for all the individuals, and for subgroups of individuals. Statistical tests will be carried out for exploratory purposes, as appropriate. The descriptive analysis of nominal/ordinal data will comprise tabulation of frequency and percentages. Chi-square test (or Fisher exact test in the presence of small frequencies) will be used to compare categories. The descriptive analysis of continuous data will comprise the mean, standard deviation, median, extreme values, and 95% confidence interval. OHS patients will be randomized to receive a short term supplementation of PRFs or placebo (J Nutr 2008), following the scheme of a controlled randomised double-blind clinical trial. POAF occurence will be compared in PRFs supplemented and control groups to assess the efficacy and safety of the intervention. The "intention to treat" principle will be adopted for the analysis of the combined endpoints.

ELIGIBILITY:
Inclusion Criteria:

* presence of sinus rhythm on the screening electrocardiogram
* first-time elective open heart surgery

Exclusion Criteria:

* absence of sinus rhythm at screening
* known allergy or intolerance to gluten or anthocyanin compound
* regularly consuming of anthocyanin or antioxidant supplements,
* being currently pregnant,
* existing or planned cardiac transplant or use of ventricular assist device,
* being unable or unwilling to provide informed consent,
* history of hepatic or renal disease,
* history of cancer history of substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Post Operative Atrial Fibrillation | up to 10 days after cardiac surgery
  Reduction of Post Operative Atrial Fibrillation after a cardiac surgery

SECONDARY OUTCOMES:
intensive unit and post-operative hospital-stay | up to hospital discharge (average period 10 days)
  reduction of intensive unit and post-operative hospital-stay
cumulative post-operative complications | up to 30 days after cardiac surgery
  reduction of occurrence of cumulative post-operative complications (renal failure, pulmonary failure (time frame: up to hospital discharge); fatal and non-fatal cardiovascular events and all-causes mortality) (time frame: up to 30 days after cardiac surgery)
circulating inflammatory markers | up to 24 hours after cardiac surgery
  additional end-point will be circulating inflammatory markers such as C reactive protein (CRP), interleukin 6 (IL6), D-dimers, plasma proteome

CONTACTS AND LOCATIONS:
Overall Officials: Licia Iacoviello, MD, PhD, Principal Investigator — IRCCS INM Neuromed, Department of Epidemiology and Prevention
Locations (1):
- IRCCS INM Neuromed, Department of Epidemiology and Prevention, Pozzilli, IS, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Costanzo S, di Niro V, Di Castelnuovo A, Gianfagna F, Donati MB, de Gaetano G, Iacoviello L. Prevention of postoperative atrial fibrillation in open heart surgery patients by preoperative supplementation of n-3 polyunsaturated fatty acids: an updated meta-analysis. J Thorac Cardiovasc Surg. 2013 Oct;146(4):906-11. doi: 10.1016/j.jtcvs.2013.03.015. Epub 2013 Apr 12. PMID 23587470